CLINICAL TRIAL: NCT07086534
Title: A Clinical Study of GeminiOne Transcatheter Edge-to-Edge Repair (TEER) System for the Treatment of Severe, Symptomatic Mitral Regurgitation (MR).
Brief Title: A Clinical Study of GeminiOne TEER System for the Treatment of Severe, Symptomatic MR.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Valve LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFSGemini1US
Record Dates: First submitted 2025-07-15; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subjects receiving the treatment of GeminiOne TEER system (Experimental)
  Interventions: Device: GeminiOne Transcatheter Edge-to-Edge Repair (TEER) System

INTERVENTIONS:
Device: GeminiOne Transcatheter Edge-to-Edge Repair (TEER) System — The GeminiOne TEER System consists of a TEER clip implant, transcatheter delivery system and a guide sheath.
  The clip is made of cobalt-chromium-nickel alloy with a nickel-titanium alloy gripper, covered with a braided mesh of polyethylene terephthalate (PET) materials.

SUMMARY:
To confirm the effectiveness and safety of the GeminiOne Transcatheter Mitral Valve Repair System for the treatment of severe, symptomatic mitral regurgitation.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, non-randomized clinical trial. All enrolled subjects will receive the investigational GeminiOne TEER System in a single-arm design. The trial will be conducted at up to seven clinical centers located in the United States, Canada, and Europe.

The GeminiOne TEER System is intended for use in adult patients with severe symptomatic mitral regurgitation (MR) who have suitable anatomy for both device implantation and transfemoral trans-septal access for left atrial delivery.

Key Inclusion Criteria:

Primary MR: Patients must be deemed high-risk for surgical intervention by the site's heart team.

Secondary MR: Patients must have failed to respond to optimal guideline-directed medical therapy (GDMT) for at least one month, and must also have received appropriate coronary revascularization and cardiac resynchronization therapy (CRT), if indicated.

Initially, up to 15 subjects will be treated. The total duration of the study is expected to be approximately 72 months. The enrollment period will span approximately 12 months. Subjects who receive the investigational device will be followed for 60 months post-implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older(≥ 18 years)
2. Subject has severe MR (Grade lll or greater per the ASE criteria, which includes severity grades of 3+ and 4+). Severity grades (3+)/ (4+) MR confirmed by core lab review on transthoracic or transesophageal echocardiography.

   For patients with primary mitral regurgitation: Deemed high or prohibitive surgical risk (STS score 8 for valve replacement or > 6 for valve repair or determined by the site heart team due to documented surgical risk factors) For patients with secondary mitral regurgitation: undergone optimal guideline-directed medical therapy (GDMT) for at least one month as determined by the local heart team; coronary revascularization, and cardiac resynchronization therapy (CRT) if clinically indicated, all of which have proven to be ineffective. Local heart team has determined that mitral valve surgery is not an option.
3. Anatomically suitable for TEER with GeminiOne device as confirmed by site investigators, core lab, and eligibility committee.
4. Feasible transseptal catheterization and femoral vein access.
5. Written informed consent from subject or legal representative.

Exclusion Criteria:

1. History of heart transplantation, prior mitral valve replacement surgery, or transcatheter mitral valve procedure.
2. Leaflet anatomy that precludes optimal positioning of the GeminiOne device, as determined by site investigators, core lab, and eligibility committee.
3. Evidence of severe calcification or significant cleft in the grasping area of the mitral valve leaflets.
4. Left ventricular ejection fraction (LVEF)< 20%
5. Left ventricular end-systolic diameter(LVESD)> 60mm
6. Mobile leaflet length less than 10mm
7. Mitral valve effective orifice area (EOA) < 3.5cm or a high risk of mitral stenosis developing after device implantation, as judged by site investigators, core lab, and eligibility committee.
8. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
9. Presence of severe non-mitral valve disease requiring intervention.
10. Severe pulmonary artery hypertension(sPAP >70mmHg).
11. Severe right ventricular dysfunction. 12, Active endocarditis or history of mitral valve endocarditis. Active rheumatic heart disease or leaflets severely degenerated from rheumatic disease.

13. Severe untreated coronary artery stenosis requiring revascularization or other cardiovascular disease requiring surgery.

14.Patents with extreme frailty. 15.Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure besides dilated cardiomyopathy.

16. Severe renal insufficiency with estimated glomerular filtration rate (eGFR) < 25 mL/min.

17. Blood cachexia including granulocytopenia(WBC<3x10^9/L),acute anemia(HB <90g/L)thrombocytopenia (PLT <50x10^9/L), severe coagulopathy, or contraindications to anticoagulant and antiplatelet therapy.

18. Evidence of an acute myocardial infarction within the past 4 weeks. 19.Evidence of stroke within the prior 90 days. 20. Any percutaneous cardiac intervention, carotid surgery, or any cardiac surgery within 30 days prior to procedure.

21. Severe symptomatic carotid artery stenosis exceeding 70% confirmed by imaging.

22. Subjects with underlying medical or psychiatric conditions that may interfere with trial evaluation (e.g. cancer, infection, severe metabolic disease). Additionally, any case deemed unsuitable for the study by the local heart team.

23.Life expectancy of less than 12 months. 24. Participation in another investigational drug or device study within the past 1 month.

25. Subjects deemed unlikely to complete the trial due to potential non-compliance, as judged by the investigator.

26. Any anatomic characteristic or presence of atrial septal occluders, which would preclude the performance of the transseptal approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety: Absence of device or procedure related major adverse events at 30 days | 30 days
  MAE is defined as the occurrence of any of the following within 30 days: death, myocardial infarction (Ml) stroke, MVARC-defined Grade 3 Acute Kidney Injury (AKl), major access site and vascular complications, major cardiac structural complications or cardiac surgery due to GeminiOne device failure.
Effectiveness: Acute procedural success (APS) | 30 days
  APS is defined as the successful implantation of the GeminiOne device and achieving residual MR of 2+ or less at discharge. lf the discharge echocardiogram is unavailable or difficult to interpret, an echocardiogram taken at 30 days can be used instead. A death before discharge or a reoperation of the mitral valve within 30 days is considered an acute procedural failure.

SECONDARY OUTCOMES:
All-cause mortality and stroke | 30 days, 12 months and annually thereafter
Cardiovascular mortality | 30 days, 12 months and annually thereafter
Rate of cardiovascular rehospitalization | 30 days, 12 months and annually thereafter
Mitral valve surgery or re-intervention | 30 days, 12 months and annually thereafter
Change in NYHA functional class | 30 days, 12 months and annually thereafter
Mitral valve hemodynamics | 30 days, 12 months and annually thereafter
  Includes degree of residual mitral regurgitation and mean mitral valve gradient.
Change in 6-Minute Walk Test (6MWT) performance | 30 days, 12 months and annually thereafter
Change in Quality of Life as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) | 30 days, 12 months and annually thereafter
Incidence of serious adverse events (SAEs) | 12 months
  A SAE is defined as any adverse event that meets one or more of the following criteria:<
  1. Death
  2. life-threatening or results in serious illness or injury
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent or significant disability/incapacity
  5. Results in a congenital anomaly/birth defect, fetal death, or fetal distress
  6. Requires medical or surgical intervention to prevent permanent impairment to a body structure or body function
  7. considered an important medical event that may jeopardize the patient or subject and/or may require intervention to prevent one of the outcomes listed above, based on appropriate medical judgment.

OTHER OUTCOMES:
Technical success | at exit from procedure room
  Must meet all of the following criteria:
  1. No procedural mortality
  2. Successful access, delivery, and retrieval of the device delivery system
  3. No emergency surgery or reintervention related to the device or access procedure
Device success | 12 months
  Must meet all of the following criteria:<
  1. No procedural mortality
  2. Proper delivery and deployment of the device
  3. No unplanned surgical or interventional procedures related to the device
  4. No specific device-related technical failure or complication
  5. Improvement of mitral regurgitation without significant stenosis (MR ≤ 2+), and without associated hemolysis or thrombogenesis